CLINICAL TRIAL: NCT05452317
Title: A Retrospective, Chart Review Study to Assess Burden of Disease Among Kidney Transplant Recipients With Chronic Active Antibody Mediated Rejection in the UK
Brief Title: Assess Burden of Disease Among Kidney Transplant Recipients With Chronic Active Antibody Mediated Rejection
Status: Completed | Type: Observational
Sponsor: CSL Behring (Industry)
Collaborators: UBC Late Stage (UK) Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: AMR BoD Study
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Antibody-mediated Rejection in Kidney Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic active AMR group
  Interventions: Other: Chronic active AMR group
- Non-Chronic active AMR group
  Interventions: Other: Non-Chronic active AMR group

INTERVENTIONS:
Other: Chronic active AMR group — Past kidney transplant. This is a retrospective, non-interventional, observational study. No study treatment will be administered in this study.
  Groups: Chronic active AMR group
Other: Non-Chronic active AMR group — Past kidney transplant. This is a retrospective, non-interventional, observational study. No study treatment will be administered in this study.
  Groups: Non-Chronic active AMR group

SUMMARY:
This study investigates the burden of disease among kidney transplant recipients that have developed Chronic Active Antibody Mediated Rejection (caAMR) compared with kidney transplant recipients that have not developed caAMR

ELIGIBILITY:
Inclusion Criteria:

Chronic Active AMR group:

* 18 Years and older
* Recipient of blood group system (ABO) compatible solitary kidney transplant between [1Jan2013] and [1Jan2018]
* Chronic active AMR diagnosed via kidney biopsy based upon Banff criteria. Patients who additionally have diagnoses such as TCMR, acute tubular necrosis, recurrence of primary kidney disease are also eligible if not the predominant pathology.
* DSA antibodies within prior 6 months of the biopsy which confirmed chronic active AMR
* Minimum of 3 years of follow up data following diagnosis of chronic active AMR (unless patient had died)
* eGFR at time of diagnosis of chronic active AMR of >25ml/min/1.73m2

Non-Chronic active AMR group:

* Age 18 years or older
* Recipient of ABO compatible solitary kidney transplant between [1 Jan 2013] and [1Jan2018]
* No documented diagnosis of chronic active AMR during the data extraction period. Patients with other diagnoses such as TCMR, acute tubular necrosis, recurrence of primary kidney disease are also eligible. Patients may or may not have had biopsies.
* Minimum of 4 years of follow up data since transplant (unless patient has died)
* eGFR of >25ml/min/1.73m2 at time of matching

Exclusion Criteria:

Chronic active AMR group:

* Recipient of a multi-organ transplant
* ABO-incompatible transplant
* Patient lost to follow up within the first 3 years post-diagnosis of chronic active AMR and whose allograft status (graft failure or patient death) is unknown.

Non-Chronic active AMR group:

* Recipient of a multi-organ transplant
* ABO-incompatible transplant
* Patient lost to follow up within the first 4 years of transplant and whose allograft status (graft failure or patient death) is unknown.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recipients of blood group system (ABO) compatible solitary kidney transplant between [1Jan2013] and [1Jan2018].
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Death censored graft loss | 5 weeks
  * eGFR<15ml/min/1.73m2 for > 60 days
  * Hemodialysis for > 60 days
  * Nephrectomy
  * Re-transplant
Decline in eGFR value over time | 5 weeks
Number of sessions received of Haemodialysis/Peritoneal Dialysis | 5 weeks
Number of patients receiving Nephrectomy | 5 weeks
Number of patients receiving re-transplantation | 5 weeks
Number of Hospital admissions per year overall | 5 weeks
Duration of hospital stay (including ICU) per year overall and by primary ICD-10 (ICD-9)/OPCS/HRG code | 5 weeks
Number of ICD-10 (ICD-9)/OPCS/HRG codes | 5 weeks
Number of A&E visits per year overall and by ICD-10 (ICD-9)/OPCS/HRG code | 5 weeks
Number of Outpatient visits per year overall and by ICD-10 (ICD-9)/OPCS/HRG code | 5 weeks
Duration and extent of Haemodialysis/Peritoneal dialysis per year | 5 weeks
Number of Treatments administered for chronic active AMR | 5 weeks
Cost of Hospital admissions (including ICU) per year overall and by ICD-10 (ICD-9)/OPCS/HRG | 5 weeks
Cost of A&E visits per year overall and by ICD-10(ICD-9)/OPCS/HRG | 5 weeks
Cost of Outpatient visits per year overall and by ICD-10 (ICD-9)/OPCS/HRG | 5 weeks
Cost of Treatment administered for chronic active AMR per year | 5 weeks
Cost of re-starting Haemodialysis/Peritoneal dialysis per year | 5 weeks
Cost of nephrectomy | 5 weeks
Cost of re-transplantations | 5 weeks

SECONDARY OUTCOMES:
Per year composite of Myocardial Infarction, Coronary revascularization, Stroke, Hospitalisation due to heart failure, and All-cause mortality | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Songkai Yan, Study Director — CSL Behring
Locations (3):
- United States (3):
  - Keck Medical Center of USC, Los Angeles, California
  - University of Maryland School of Medicine, Div. of Nephrology, Baltimore, Maryland
  - The Washington University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No